CLINICAL TRIAL: NCT01042444
Title: Phase I Study to Demonstrate the Safety and Performance of the GARDEX™ Embolic Protection Device When Used During Percutaneous Coronary Intervention (PCI) of Saphenous Vein Graft
Brief Title: Use of the GARDEX™ Embolic Protection Device During Percutaneous Coronary Interventions of Saphenous Vein Graft
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Gardia Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gardia Medical Ltd.
Record Dates: First submitted 2009-12-30; First posted 2010-01-05 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Saphenous Vein Graft Disease; Myocardial Ischemia; Embolism
Keywords: Heart disease; Embolic Protection Device; PCI; SVG
MeSH Terms: conditions — Myocardial Ischemia; Embolism; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Embolic Protection Device (Experimental): The study will involve up to 20 patients to be enrolled using the GARDEX system during clinically indicated percutaneous intervention of SVG and followed through 30 days post procedure. Patients will be enrolled at up to 3 investigative sites. The study is a prospective multi center registry with sequential enrollment of qualified patients who consent to participate and meet the eligibility criteria.
  Interventions: Device: GARDEX™

INTERVENTIONS:
Device: GARDEX™ — GARDEX is an embolic protection system to contain and remove embolic material (thrombus/debris) during cardiovascular interventions.
  The diameter of the vessel at the site of filter basket placement should be between 3.5 mm to 6.0 mm. The GARDEX Embolic Protection System may be used with commercially available 0.014" guide wires.

SUMMARY:
This is a multi center, prospective study designed to demonstrate the safety and performance of the GARDEX Embolic Protection System when used as an adjunctive device during saphenous vein graft (SVG) interventions.

ELIGIBILITY:
Inclusion Criteria:

* Anticipated patient life expectancy of at least 1 year from enrollment.
* Patient (or their legal guardian) has provided a signed informed consent.
* Patient is willing to comply with the protocol requirements.
* Candidate for PCI, stenting and CABG.
* Total CK verified to be within hospital normal limits at the time of enrollment.
* Myocardial ischemia as evidenced by one or more of the following:

  * Diagnosis at time of enrollment of stable or unstable angina pectoris
  * Reversible 12 lead ECG changes consisted with ischemia
  * Positive function study (e.g. stress test)
  * Recent myocardial infarction (>24 hours prior to enrollment with total CK verified to be within hospital normal limits at the time of enrollment).
* Lesions amendable to PCI.
* Lesion(s) is located within SVG and has ≥50% and <100% stenosis (angiographic visual assessment).
* Only single SVG graft to be treated.
* Vessel has thrombolysis in myocardial infarction (TIMI) grade 1 or higher flow before the passage of a guidewire.
* Reference vessel diameter where the GARDEX™ system is to be placed is ≥ 3.5mm and ≤6.0mm in diameter by angiographic visual estimation.

Exclusion Criteria:

* A hypersensitivity or contraindication to heparin and bivalirum (Angiomax), aspirin, ticlopidine, clopidogrel, murine products, procedure equipment material, and a sensitivity to contrast dye which cannot be adequately pre-treated with diphenhydramine and/or steroids.
* Myocardial infarction with documented total CK> 2 times the upper limit of normal within the past 24 hours, or currently experiencing an acute myocardial infarction.
* A stroke or transient ischemic attach (TIA) within the past 2 months.
* A history of bleeding diathesis or coagulopathy.
* Major gastrointestinal (GI) bleeding within 3 months of index procedure.
* Baseline creatinine ≥ 2.5 mg/dl.
* A planned invasive surgical procedure within 30 days.
* Undergone cardiac surgery within the past 60 days.
* The lesion is in a SVG that is less than 2 months post implant.
* Left ventricular ejection fraction < 20%
* The lesion is an arterial conduit.
* Anatomical exclusions that preclude placement of the GARDEX™ system per the Instruction for Use.
* More than one SVG graft that need to be treated at the index procedure.
* Chronic occlusion of the target lesion/severe calcification.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the safety and performance of the GARDEX Protection System. The primary end point is the combined rate of major adverse events (MACE) at 30 days. | 30 days

SECONDARY OUTCOMES:
The secondary study objectives includes Device,Angiographic,Procedural and Clinical Success ,Final TIMI flow grade, Angiographically evident emboli | Device,Angiographic, Procedural Success ,Final TIMI flow grade, Angiographically evident emboli-Procedural; Clinical Success-30 days

CONTACTS AND LOCATIONS:
Overall Officials: Uri Rosenschein, MD, Principal Investigator — Bnei Zion Hospital, Haifa Israel
Locations (3):
- Israel (3):
  - Bnai Zion Medical Center, Haifa
  - Rabin Medical Center - Beilinson Campus, Petah Tikva
  - Tel-Aviv Sourasky Medical Center, Ichilov Hospital, Tel Aviv